CLINICAL TRIAL: NCT04307927
Title: Lifetech LAmbre™ Left Atrial Appendage Closure System Post-Market Registry Single-center, Single-arm, Prospective, Post-market Registry
Brief Title: Lifetech LAmbre™ Left Atrial Appendage Closure System Post-Market Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LA-PMCF-02
Record Dates: First submitted 2020-03-12; First posted 2020-03-13 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Atrial Fibrillation
Keywords: Left atrial appendage occluder
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single-center, single-arm, prospective, post-market study of LAmbre™ LAA Closure System. To evaluate immediate and long term procedural success of Lifetech LAmbre™ occluders in patients.

DETAILED DESCRIPTION:
Detailed Description:

Atrial fibrillation (AF) is the most common cardiac arrhythmia causing ischemic stroke. The CHA2DS2-VASc score was developed to estimate the stroke rate in patients with non-valvular AF, and high scores predict a raised annual stroke risk. The yearly stroke risks without treatment in patients with CHA2DS2-VASc score 2 and 9 are 2.2% and 15.2% respectively. For patients with increased stroke risk (CHA2DS2-VASc score ≧2), warfarin or other novel oral anticoagulants (NOAC) recommended for stroke prevention. Despite the effectiveness of current pharmacological therapies for stroke prevention in atrial fibrillation, around 20% of patients discontinue therapy - whether new oral anticoagulants (NOAC) or warfarin because of side effects and/or bleeding. In addition, warfarin needs to be dosed individually to target an international normalized ratio (INR) of 2-3 for striking an optimal balance between bleeding and ischemic stroke events. This, combined with drug-drug interaction that occurs with both NOACs and warfarin, results in inadequate stroke protection in a substantial portion of AF patients. The LAA is the source of 90% of cardiac emboli attributed to stroke events. This is a windsock-like structure on the lateral border of the left atrium with internal trabeculations, and being a confined space, is prone to blood stasis and thrombus formation. Currently, there are surgical, epicardial and percutaneous techniques for occluding this structure in order to reduce stroke in AF patients cannot take long term oral anticoagulants, and the percutaneous route is intuitively the most attractive given its relative non-invasiveness. The two devices in most widespread use for percutaneous LAA closure worldwide are the Watchman (Boston Scientific, Natick, MA, USA) and the Amplatzer Cardiac Plug (ACP) (Abbott, IL, CA USA). However, both devices have limitations including the need for relatively large delivery sheaths (9-14 French) and limited recapture and repositioning capabilities.

LAmbreTM LAA Closure System (Lifetech Scientific, Shenzhen, China) is a novel self-expanding LAA occluder constructed from a nitinol mesh and polyester membranes and consists of an umbrella and a cover connected by a short central waist. The device is delivered by an 8-10 French sheath and has full recapture and repositioning capabilities. LAmbreTM LAA Closure System received the CE mark in June 2016.

This PMCF study will be carried out following the CE mark of LAmbreTM LAA Closure System and is intended to confirm the effectiveness and safety of LAmbreTM LAA Closure System.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must be at least 18 years of age; 2. Patients with non-valvular paroxysmal, persistent or permanent atrial fibrillation with long-term sustainability scheduled for interventional LAA closure; 3. Patient characteristics consistent with the corresponding IFU and sizing guidelines*; 4. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Ethics Committee (EC); 5. The patient agrees to comply with requirements of the study including the 24 months follow- up.

Exclusion Criteria:

* 1. Any contra-indication mentioned in the corresponding IFU*; 2. Currently participating in other investigational drug- or device studies; 3. Patient who is pregnant, planning to become pregnant, or breast feeding; 4. Patients cannot tolerate transoesophageal echocardiogram (TEE).

  * Note: In IFU, the Left Atrial Appendage Closure System is contraindicated for the following: • Patients' LAA anatomy not suitable for the REF of the device.

    * Patients' with intracardiac thrombus.
    * Patients with active endocarditis or other infections causing bacteremia.
    * Patients where placement of the device would interfere with any intracardiac or intravascular structures.
    * Patients with contraindications to X-Ray and/or trans-esophageal echocardiographic examinations.
    * Patients with known hypersensitivity to nickel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular paroxymal, persistent or permanent atrial fibrillation with long-term sustainability scheduled for interventional LAA closure.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1.Absence of peri-procedural stroke/TIA, device embolization, cardiac or vascular perforation, any other device or procedure related serious adverse event or death (procedure or device related or of unknown cause); | 7 days
  Peri-procedure defined as within 7 days of the procedure.
Implant success | 1 day
  Implant success defined as correct positioning and release of the occluder device into the proper anatomical location. Correct positioning is assessed as absence of major residual jet flow (>5mm) into the LAA closure with the device evaluated by transesophageal echocardiogram (TEE).

SECONDARY OUTCOMES:
Incidence of stroke or systemic embolism or death through 24 months post implantation | 24 months
  Incidence of stroke or systemic embolism or death through 24 months post
Successful sealing around the device at the LAA orifice with residual jet ≤5 mm flow measured by TEE at 1-3 months, 6 months post-implantation | 1-3 months, 6 months post-implantation
  Successful sealing around the device at the LAA orifice with residual jet ≤5 mm flow measured by TEE at 1-3 months, 6 months post-implantation
Device or procedure related Serious Adverse Events (SAEs) from attempted procedure through 24 months post implantation | 24 months
  Device or procedure related Serious Adverse Events (SAEs) from attempted procedure through 24 months post implantation
All SAEs (death included) from attempted procedure through 24 months post implantation | 24 months
  All SAEs (death included) from attempted procedure through 24 months post implantation
Incidence of bleeding event through 24 months post implantation. | 24 months
  Incidence of bleeding event through 24 months post implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangtao Yu, Professor, Principal Investigator — Katholisches Klinikum Koblenz ·Montabaur
Locations (1):
- Katholisches Klinikum Koblenz ·Montabaur, Koblenz, Germany